CLINICAL TRIAL: NCT02382055
Title: Changing Habits in Anorexia Nervosa
Brief Title: Changing Habits in Anorexia Nervosa: Novel Treatment Development
Acronym: REACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7072
Record Dates: First submitted 2015-01-29; First posted 2015-03-06 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Anorexia Nervosa
Keywords: Eating Disorders; Psychotherapy; Anorexia Nervosa; Treatment
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- REACH (Experimental): Psychotherapy
  Interventions: Behavioral: REACH; Behavioral: Inpatient Behavioral Treatment
- Supportive Psychotherapy (Active Comparator): Psychotherapy
  Interventions: Behavioral: Supportive Psychotherapy; Behavioral: Inpatient Behavioral Treatment

INTERVENTIONS:
Behavioral: REACH — REACH is a 12-session intervention, delivered 2-3 times per week for 45 minutes. The treatment focuses on identifying and changing behaviors and routines that have become entrenched and help perpetuate the illness.
  Arms: REACH
Behavioral: Supportive Psychotherapy — The Supportive Psychotherapy is based on the Specialist Supportive Care (McIntosh et al, 2005), and modified for the current research procedures. Supportive Psychotherapy is a 12-session intervention, delivered 2-3 times per week as 45 minute sessions, focusing on symptoms of anorexia nervosa during the transition to the inpatient unit.
  Arms: Supportive Psychotherapy
Behavioral: Inpatient Behavioral Treatment — Inpatient treatment at the NYSPI is a behaviorally-based treatment program for anorexia nervosa. This is a non-research, clinical intervention for individuals with anorexia nervosa.

SUMMARY:
The investigators are examining what types of psychotherapy are most helpful for patients as they undergo weight restoration treatment for anorexia nervosa. In this study, patients who are receiving care on our inpatient unit will also receive 4 weeks of one two types of psychotherapy: Supportive Psychotherapy or Regulation Emotions and Changing Habits.

DETAILED DESCRIPTION:
Patients will be receiving specialized inpatient treatment for anorexia nervosa on the Eating Disorders Unit at the New York State Psychiatric Institute, where care is provided free of charge.

Study procedures will begin after one week of acclimating to the inpatient unit. Patients will be randomly assigned to receive either Supportive Psychotherapy (focused on the transition to the inpatient unit) or REACH (focused on changing routines or habits that have become part of the eating disorder). Each treatment consists of 12-sessions, delivered 2-3 times per week.

Before and after treatment, patients will be asked to participate in interviews, questionnaires, and a lunch meal.

ELIGIBILITY:
Inclusion Criteria:

* DSM5 diagnosis of anorexia nervosa
* Age>= 18
* Medically stable
* Able to provide informed consent

Exclusion Criteria:

* Other psychiatric disorder requiring acute treatment
* Serious medical illness
* Antipsychotic medication
* Severe cognitive impairment

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Habit strength as measured by self report scales | 4 weeks

SECONDARY OUTCOMES:
Eating behavior as measured by laboratory meal | 4 weeks
Eating behavior as measured by meal observation | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Steinglass, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Background] Foerde K, Knowlton BJ, Poldrack RA. Modulation of competing memory systems by distraction. Proc Natl Acad Sci U S A. 2006 Aug 1;103(31):11778-83. doi: 10.1073/pnas.0602659103. Epub 2006 Jul 25. PMID 16868087
- [Background] McIntosh VV, Jordan J, Carter FA, Luty SE, McKenzie JM, Bulik CM, Frampton CM, Joyce PR. Three psychotherapies for anorexia nervosa: a randomized, controlled trial. Am J Psychiatry. 2005 Apr;162(4):741-7. doi: 10.1176/appi.ajp.162.4.741. PMID 15800147
- [Background] McGowan L, Cooke LJ, Gardner B, Beeken RJ, Croker H, Wardle J. Healthy feeding habits: efficacy results from a cluster-randomized, controlled exploratory trial of a novel, habit-based intervention with parents. Am J Clin Nutr. 2013 Sep;98(3):769-77. doi: 10.3945/ajcn.112.052159. Epub 2013 Jul 17. PMID 23864536
- [Background] Walsh BT. The enigmatic persistence of anorexia nervosa. Am J Psychiatry. 2013 May;170(5):477-84. doi: 10.1176/appi.ajp.2012.12081074. PMID 23429750